CLINICAL TRIAL: NCT04644419
Title: Chemotherapy-related Cognitive Impairment in Adults With Acute Leukemia
Brief Title: Chemotherapy-related Cognitive Impairment and Acute Leukemia
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2045
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Cognitive function
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control group of the LCCC1848: Patients in the control arm will receive standard of care.
  Interventions: Other: none (observational study)

INTERVENTIONS:
Other: none (observational study) — This is an observational study and does not include intervention delivery.

SUMMARY:
This is an ancillary study of an intervention study (NCT04570709). The parent study is a single institution, feasibility trial of 20 (10 control and 10 intervention) patients with the primary objective of assessing feasibility, acceptability, and change in pre and post measures of symptoms, function, and quality of life by administering the Palliative and Collaborative Care InTervention (PACT). We will further assess cognitive function in the patients who participate in the control of the parent study.

DETAILED DESCRIPTION:
The study objective is to observe patient-reported and researcher-assessed cognitive function in adults with acute myeloid leukemia with chemotherapy treatment. We will assess cognitive function using a battery of neuropsychological assessments, patient-reported questionnaire, and semi-structured interviews among participants in control group only. The group assignment will be conducted through parent study (NCT04570709). Participating in this study will not affect participants' group assignment.

ELIGIBILITY:
[Patient]

Inclusion Criteria:

* ≥ 60 years of age
* diagnosis of AML
* Receive 1) low-dose cytarabine or hypomethylating agent (HMA) in combination with Venetoclax chemotherapy OR 2) low-dose cytarabine or hypomethylating agent (HMA) in combination with Venetoclax chemotherapy and any investigational drugs
* have caregiver(s) willing to participate
* participate in the parent study (PACT study, NCT04570709)

Exclusion Criteria:

* referred to hospice care

[Caregiver]

Inclusion criteria:

* identified by patient as a caregiver
* ≥18 years of age
* speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years or older, diagnosed with AML, received HMA+VEN treatment, and participated in the NCT04570709 study.
  Caregivers identified by eligible patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Cognitive function as assessed by Functional Assessment of Cancer Therapy - Cognitive Function | at the second cycle of treatment (about day 30)
  The questionnaire consists of 4 domains, including perceived cognitive impairments, comments from others, perceived cognitive abilities, and impact of quality of life. The higher the score, the better the cognitive function.
Processing speed and executive function as assessed by Trial Making Test | at the second cycle of treatment (about day 30)
  Include both trails A and B.
Memory and verbal learning as assessed by Hopkins Verbal Learning Test-revised (HVLT-R) | at the second cycle of treatment (about day 30)
  Include total recall and delayed recall.
Speeded lexical fluency as assessed by Delis-Kaplan Executive Function System (D-KEFS) letter fluency | at the second cycle of treatment (about day 30)
  Include three initial alphabet letter for each assessment.
Attention and working memory as assessed by Wechsler Adult Intelligence Scale (WAIS)-digit span | at the second cycle of treatment (about day 30)
  Include forward and backward assessment.
Cognitive effort as assessed by Borg CR 10 | at the second cycle of treatment (about day 30)
  Range from 0-10, maximum. The higher the score, the much the cognitive effort.

SECONDARY OUTCOMES:
Cognitive function as assessed by Functional Assessment of Cancer Therapy - Cognitive Function | at the first, third, fourth, fifth, sixth, and seventh cycle of treatment (baseline, about day 60, 90, 120, 150, and 180)
  The questionnaire consists of 4 domains, including perceived cognitive impairments, comments from others, perceived cognitive abilities, and impact of quality of life. The higher the score, the better the cognitive function.
Processing speed and executive function as assessed by Trial Making Test | at the first, fourth, and seventh cycle of treatment (baseline, about day 90 and 180)
  Include both trails A and B.
Memory and verbal learning as assessed by Hopkins Verbal Learning Test-revised (HVLT-R) | at the first, fourth, and seventh cycle of treatment (baseline, about day 90 and 180)
  Include total recall and delayed recall.
Speeded lexical fluency as assessed by Delis-Kaplan Executive Function System (D-KEFS) letter fluency | at the first, fourth, and seventh cycle of treatment (baseline, about day 90 and 180)
  Include three initial alphabet letter for each assessment.
Attention and working memory as assessed by Wechsler Adult Intelligence Scale (WAIS)-digit span | at the first, fourth, and seventh cycle of treatment (baseline, about day 90 and 180)
  Include forward and backward assessment.
Cognitive effort as assessed by Borg CR 10 | at the first, fourth, and seventh cycle of treatment (baseline, about day 90 and 180)
  Range from 0-10, maximum. The higher the score, the much the cognitive effort.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ning Chan, MSN, RN, Principal Investigator — University of North Carolina, Chapel Hill; Ashley L Bryant, PhD, RN, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehenisive Cancer Center, Chapel Hill, North Carolina, United States